CLINICAL TRIAL: NCT02846233
Title: Is the Stepping-down Approach a Better Option Than Multiple Daily Injections in Patients With Chronic Poorly-controlled Diabetes on Advanced Insulin Therapy?
Brief Title: Stepping-down Approach in Patients With Chronic Poorly-controlled Diabetes on Advanced Insulin Therapy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDMSTEP
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; dulaglutide; Insulin Glargine; Insulin Detemir; Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Interventions: All prandial insulin injections, usually 3 times daily before meals, will be discontinued. Basal insulin, usually once daily at bed time, will be continued at 80 % of the home dose. Albiglutide OR Dulaglutide AND Empagliflozin will be added to metformin and a basal insulin.
  Interventions: Drug: GLP1 receptor agonist; Drug: basal insulin; Drug: SGLT2 inhibitor; Drug: Metformin
- Control group (No Intervention): Interventions: There will not be any change in insulin therapy, and they will continue to have the usual and standard care through the primary care provider. They should not receive SGLT2i and GLP1 RA during the study period.

INTERVENTIONS:
Drug: GLP1 receptor agonist — "Albiglutide or Dulaglutide" will be added to a basal insulin.
  Other Names: Albiglutide (Tanzeum) or , Dulaglutide (Trulicity)
  Arms: Treatment group
Drug: basal insulin — The participant will continue with the basal insulin.
  Other Names: Lantus, Toujeo, NPH, levemir
  Arms: Treatment group
Drug: SGLT2 inhibitor — "Empagliflozin" will be added to a basal insulin.
  Other Names: Empagliflozin (Jardiance)
  Arms: Treatment group
Drug: Metformin — The participant will continue with metformin.
  Arms: Treatment group

SUMMARY:
In traditional step-up approach, the patients with poorly-controlled type 2 diabetes are instructed to take up to 4 insulin injections daily or multiple daily injections (MDI) as the most advanced therapy. However, a significant number of these patients continue to have poor diabetes control. The most common reason is the noncompliance with multiple injections and the patient's reluctance to accept insulin-induced weight gain. More recently, the algorithm in diabetes management has significantly changed to accommodate the newer generation of medications. Addition of the diabetes medications, that can induce weight loss such as oral Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors and once-weekly glucagon-like peptide (GLP)-1 receptor agonists (GLP1 RA) injection, to a basal insulin is now recommended before the patient is advanced to MDI. This approach works very well in most patients since weight loss gives the patients an extra motivation to take medication regularly. Similarly, the patient does not require to take an insulin injection before each meal throughout the day in this approach.

Unfortunately, there are still a large number of patients with poor glycemic control who are still on MDI. Some of them were initiated on MDI before the availability of newer generations of medications. Some were started simply because the physician was not aware of or not the familiar with the new recommendations. Regardless of the reason, these patients are likely to remain on MDI despite chronic poor glycemic control since the physicians are understandably reluctant to step down the most advanced insulin therapy. In addition, there has been no data on the benefits and safety of the stepping-down approach from the most advanced insulin therapy to the more patient-friendly approach that is the combined use of oral SGLT2i and once-weekly GLP1 RA injection.

DETAILED DESCRIPTION:
A prospective, randomized, open-label, controlled, parallel-group trial is planned. This study is an interdepartmental collaborative study among the Department of Internal Medicine, Department of Family & Community Medicine (UCSF Fresno), Sierra Vista Family Medicine Residency Program and Division of Endocrinology.

The study will be conducted at the following multiple locations in order to maximize the patient recruitment:

1. Internal medicine clinic at Derian Koligian ambulatory care center (ACC)
2. Family practice medicine clinic at ACC
3. Diabetes clinic at ACC
4. Internal medicine clinic at University Medicine Associates in East medical Plaza
5. Endocrine clinic at University Medicine Associates in East medical Plaza
6. Sierra Vista clinics

The patients will be recruited during the first 12 months of the study or until the predetermined sample size is reached, whichever comes first.

The patient's primary care provider will be informed of the enrollment in the study if the participant gives the permission to do so.

All participants in both group will need to make all 3 visits to UCSF Clinical Research Center over 16- week period.

(1) First visit: Once the site co-investigators identify the suitable and interested study patient, a trained research coordinator will contact the patient for the first visit. The patient will be seen at the UCSF Clinical Research Center by the research coordinator and a physician co-investigator.

During the first visit, all patients in both group will

* be given the information about the study.
* sign the consent form.
* be randomly assigned to either treatment (i.e. Step Down) or control (MDI) group by using A Randomization Plan from http://www.randomization.com.
* have the blood test for A1c, CMP, CBC, fasting lipid and measurements of body weight, height, blood pressure, and heart rate.
* complete both the Diabetes Medications Satisfaction (DM-SAT) Questionnaire form and the Brief Medication Questionnaire (BMQ).

Medication changes at first visit:

In treatment group,

1. All prandial insulin injections (Humalog, Novolog, Apidra, Novolin R or Humulin R), usually 3 times daily before meals, will be discontinued.
2. Basal insulin (NPH, Lantus, Levimir, Toujeo or Tresiba), usually once daily at bed time, will be continued at 80 % of the home dose. The dose will be gradually increased until the patient is back on the home dose (the dose that the patient has been taking at home prior to the enrollment) or fasting BG of 80-130mg/dl is achieved by using the self-titration regimen.
3. If the patient is on pre-mixed basal+prandial insulin 2-3 times daily, it will be discontinued and a basal insulin alone, (NPH, Lantus, Levemir, Toujeo or Tresiba), will be given at 40% of total daily dose of pre-mixed insulin. The dose will be gradually increased until fasting BG of 80-130mg/dl is achieved by using the self-titration regimen.
4. Metformin, that most patients are expected to be on, will be continued, but other non-insulin oral medications for diabetes will be discontinued. If the patient is not on metformin, then Metformin ER will be started at 500mg with a meal for 2 weeks as a routine care and then 1000mg daily as a maintenance dose if tolerated.
5. Both SGLT2i and GLP1 RA will be added to metformin and a basal insulin.

The patient will be trained on the injection technique of the once-weekly GLP1 RA, potential side effects, risk and benefits of all new medications in detail, hypoglycemia management and the self-titration regimen for the basal insulin.

In the control group, there will not be any change in MDI therapy, and the participants will continue to have the usual and standard care through the primary care provider. The participants should not receive SGLT2i and GLP1 RA during the study period.

(2) Second visit: At 4 weeks after the patient starts taking new medications, the patients will make the 2nd visit to the UCSF Clinical Research Center.

During the 2nd visit, the patient in the treatment group will

* be enquired about any side effect of the medications.
* be reviewed on insulin dose and the use of self-titration regimen for the basal insulin.
* have the blood test for A1c, CMP, CBC, fasting lipid and measurements of body weight, height, blood pressure, and heart rate.
* complete both the Diabetes Medications Satisfaction (DM-SAT) Questionnaire form and the Brief Medication Questionnaire (BMQ).

In the control group, there will not be any change in MDI therapy, and the participants will continue to have the usual and standard care through the primary care provider. The participants should not receive SGLT2i and GLP1 RA during the study period.

During the 2nd visit, the patient in the control group will

* have the blood test for A1c, CMP, CBC, fasting lipid and measurements of body weight, height, blood pressure, and heart rate.
* complete both the Diabetes Medications Satisfaction (DM-SAT) Questionnaire form and the Brief Medication Questionnaire (BMQ).

  (3) Third visit: The patients will make the 3rd or final visit to the UCSF Clinical Research Center at 12 weeks after 2nd visit or 16 weeks from the date of the start of both SGLT2i and a GLP1 RA.

During the 3rd visit, the patients in both groups will

* have the blood test for A1c, CMP, CBC, fasting lipid and measurements of body weight, height, blood pressure, and heart rate.
* complete both the Diabetes Medications Satisfaction (DM-SAT) Questionnaire form and the Brief Medication Questionnaire (BMQ).

The investigators will try to make a clinic appointment with primary care provider one month prior to the last visit to the research center for those who are in the treatment group if the patient gives the permission to do so. Therefore the primary care provider will be able to order the medications through the patient's health insurance plan if the patient wishes to remain on the study medications beyond the study period. Alternatively, the patients can go back on insulin therapy that was given prior to the study.

Monitoring of the treatment group:

The patients in both groups will monitor FPGs daily at minimum. The research coordinator will call all participants in both groups at weeks 1, 2, 8, and 12 to review fasting glucose measurements, ask for possible adverse events, incidents of hypoglycemia, and any change in medication.

All participants in both groups in both groups will be reviewed again at the UCSF Clinical Research Center at weeks #4 and #16 for both blood tests and physical examinations.

Outcome measurements:

The primary outcome is the change in A1c at the end of 16 weeks of study period and secondary outcomes are the changes in fasting blood glucose, weight, blood pressure, heart rate, fasting lipids, serum sodium and potassium, serum creatinine, liver enzymes, CBC, medication adherence scores and treatment satisfaction scores . These changes will be compared between the two independent groups, namely the treatment group and the control group, and also within the same group.

Blood test and questionnaire:

The following blood work will be drawn and analyzed at the community regional medical center at baseline (first visit), at 4 weeks and at the end of the study at 16 weeks:

1. A1c
2. Complete Blood Count (CBC) with differential
3. Complete metabolic panel (CMP)
4. Fasting lipid profile

Patient satisfaction with treatment in both groups will be measured by the validated the Diabetes Medications Satisfaction (DM-SAT) Questionnaire form.

Patient adherence will be determined by using the Brief Medication Questionnaire (BMQ).

SAMPLE SIZE AND ANALYSIS PLAN:

The investigators will attempt to recruit and consent 20 patients in each arm that was calculated to provide an 80% statistical power at a 0.05 alpha in this continuous endpoint, two independent sample study.

The calculation was based on the following:

A mean Hemoglobin A1c of 8.5±1% at the initiation of the study period. In the treatment group we anticipate a decline in Hemoglobin A1c of 12-15% by the end of the study period. The standard deviation for the mean A1c was derived from the literature.

The data will be analyzed by using SPSS software. Significance testing will be conducted at the two-sided 5% level. Continuous variables will be examined for normality and if assumption is met, differences in mean values will be tested using Student's t test an analysis of variance (ANOVA). If not normally distributed, non-parametric procedures will be used, including Wilcoxan rank Sum test. Categorical data will be analyzed using Fisher's exact test and Chi square analysis. Since before/after comparisons will also be performed on the same study patients we will utilize paired t tests and McNemar's chi-square test.

ELIGIBILITY:
Inclusion Criteria:

The following patients with diabetes mellitus type 2 who can give written consent will be eligible for enrollment. They must meet all criteria.

1. > 21 years of age
2. Body mass index (BMI) ≥30 kg/m2
3. On insulin at least 2 times daily comprising both a basal and a prandial insulin or a pre-mix insulin with or without other non-insulin medications for a least past 3 months
4. A1c >8%
5. eGFR >45%

Exclusion Criteria:

The patients with any of the following criteria will be excluded.

1. Any patient who does not meet the above inclusion criteria.
2. Pregnancy
3. Patients who are on a SGLT2i and a GLP1 RA injection at the time of enrollment.
4. diabetes mellitus type 1
5. C-peptide below normal range if measured in the past.
6. patients with a history of diabetes ketoacidosis
7. A history of recent and frequent (≥ 2 times within past 3 months) urinary tract infection or genito-urinary candidiasis requiring antibiotic and/or anti-fungal therapies.
8. a personal or family history of medullary thyroid carcinoma (MTC) or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
9. eGFR <45%
10. patients with a history of acute pancreatitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SOE NAING, MD, Principal Investigator — UCSF - Fresno
Locations (1):
- UCSF Fresno, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman WH, Kalyani RR, Wexler DJ, Matthews DR, Inzucchi SE. Response to Comment on American Diabetes Association. Approaches to Glycemic Treatment. Sec. 7. In Standards of Medical Care in Diabetes-2016. Diabetes Care 2016;39(Suppl. 1):S52-S59. Diabetes Care. 2016 Jun;39(6):e88-9. doi: 10.2337/dci16-0003. No abstract available. PMID 27222560
- [Background] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, DeFronzo RA, Einhorn D, Fonseca VA, Garber JR, Garvey WT, Grunberger G, Handelsman Y, Henry RR, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE; American Association of Clinical Endocrinologists (AACE); American College of Endocrinology (ACE). CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM--2016 EXECUTIVE SUMMARY. Endocr Pract. 2016 Jan;22(1):84-113. doi: 10.4158/EP151126.CS. No abstract available. PMID 26731084
- [Background] Diamant M, Nauck MA, Shaginian R, Malone JK, Cleall S, Reaney M, de Vries D, Hoogwerf BJ, MacConell L, Wolffenbuttel BH; 4B Study Group. Glucagon-like peptide 1 receptor agonist or bolus insulin with optimized basal insulin in type 2 diabetes. Diabetes Care. 2014 Oct;37(10):2763-73. doi: 10.2337/dc14-0876. Epub 2014 Jul 10. PMID 25011946

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 12 | 10
Completed | 10 | 8
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Customized [Mean (Standard Deviation); unit: years] | 51.8 (11.14) | 55.65 (11.78) | 53.5 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanics | 8 | 5 | 13
  White | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c at the End of Study Period
Description: change in A1c (%) from baseline to end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: % change of A1c
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
% change of A1c | -2.38 [-2.93 to -1.83] | -0.83 [-2.05 to 0.40]

2. Secondary Outcome: Changes in Weight
Description: change (in pounds) from baseline to the end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
pounds | -16.38 [-25.63 to -7.13] | -0.1 [-1.34 to 1.14]

3. Secondary Outcome: Changes in Blood Pressure
Description: change (mmHg) of systolic BP from baseline to the end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
mmHg | -16 [-33.37 to 1.37] | 15 [2.56 to 27.44]

4. Secondary Outcome: Changes in Heart Rate
Description: change (beats/min) from baseline to the end of study at 16 weeks
Time Frame: 16 weeks
Measure: Mean (95% Confidence Interval); unit: beats per min
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
beats per min | 4.3 [-1.05 to 9.65] | 5.13 [-3.93 to 14.18]

5. Secondary Outcome: Changes in LDL
Description: change (mg/dL) from baseline to the end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
mg/dL | -15.7 [-30.29 to -1.11] | 21 [-9.9 to 51.9]

6. Secondary Outcome: Changes in Total Cholesterol
Description: change (mg/dL) from baseline to the end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
mg/dL | -18.5 [-35.79 to -1.21] | 18.38 [-22.38 to 59.13]

7. Secondary Outcome: Changes in Serum Creatinine
Description: change (mg/dL) from baseline to the end of study at 16 weeks
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
mg/dL | 0.04 [-0.08 to 0.16] | 0.04 [-0.04 to 0.11]

8. Secondary Outcome: Changes in Treatment Satisfaction Scores (DM-SAT Total Score)
Description: Patient satisfaction with treatment in both groups will be measured by the validated the Diabetes Medications Satisfaction Tool (DM-SAT). Response options range from 0="not at all satisfied" to 10="extremely satisfied" and a total score is calculated ranging from 0 to 100, with higher scores indicating more diabetes medication satisfaction.
Time Frame: 16 weeks (from baseline to end of study at 16 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 10 | 8
score on a scale | 45.3 [28.19 to 62.41] | 4.63 [-0.83 to 10.08]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 10/12 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=12) | Control Group (N=10)
Mild hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Mild hypoglycemia event (BG 40-69 mg/dL)
Nausea (Gastrointestinal disorders) | 9 (9) | 0 (0)
Severe hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Severe hypoglycemia event (BG <40 mg/dL)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02846233/Prot_SAP_000.pdf